CLINICAL TRIAL: NCT07148518
Title: Comparison of Upper and Lower Limb Maximal Exercise Capacities, Arterial Stiffness, Muscle Oxygenation and Energy Consumption During Tests in Patients With Coronary Artery Disease
Brief Title: Comparison of Upper and Lower Limb Maximal Exercise Capacities and Arterial Stiffness in Patients With CAD
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Head of Cardiopulmonary Rehabilitation Clinic, Gazi University
Other Study IDs: Gazi University 76
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: coronary artery disease; cardiopulmonary exercise testing; arterial stiffness; oxygen consumption
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lower Extremity Group: The first test is the cardiopulmonary exercise test (CPET), which evaluates the maximal exercise capacity of the lower extremities and will be performed on a treadmill. During the test, the muscle oxygen of the individuals will be measured with a near-infrared spectrometer, and their energy consumption will be measured with a multisensory physical activity monitor. Additionally, both arterial stiffness, assessed with the arteriograph device, and respiratory muscle fatigue, evaluated using a mouth pressure measurement device, will be measured before and after the test.
- Upper Extremity Group: In the second test, the maximal exercise capacity for the upper limb will again be evaluated by CPET and performed on the arm ergometer. The second test will be conducted 48 hours after the lower extremity exercise test. During the test in the second group, as in the first test, muscle oxygen will be measured with a near-infrared spectrometer, and energy expenditure with a multisensory physical activity monitor. Furthermore, arterial stiffness, determined by the arteriograph device, and respiratory muscle fatigue, assessed through a mouth pressure measurement system, will both be evaluated pre- and post-test.

SUMMARY:
Coronary artery disease (CAD) significantly increases mortality rates in both developed and developing countries. In this condition, the impairment of arterial blood circulation leads to insufficient blood supply to the myocardium during both rest and exercise, resulting in symptoms such as angina pectoris, dyspnea, and fatigue. Patients, particularly due to their fear of experiencing angina pectoris, tend to adopt a sedentary lifestyle. This situation contributes to exercise intolerance and a reduction in exercise capacity among individuals with CAD. A review of the literature reveals a lack of studies investigating upper and lower extremity exercise capacity and the physiological responses during exercise testing in patients with CAD. Therefore, the aim of this study is to compare arterial stiffness, muscle oxygenation, respiratory muscle fatigue, energy expenditure, perceived dyspnea, and fatigue during upper and lower extremity exercise testing in patients with coronary artery disease.

DETAILED DESCRIPTION:
As a consequence of atherosclerosis progresses with aging, the lumen of the arteries narrows and the arterial wall thickens. In patients with coronary artery disease, this process impairs arterial blood flow, resulting in insufficient blood supply to the myocardium. Consequently, due to the inability to meet the oxygen demands of the heart muscle both at rest and during exercise, patients experience symptoms such as angina pectoris, dyspnea, and fatigue. Particularly, fear of developing angina pectoris during physical activity leads patients to develop kinesiophobia and adopt a sedentary lifestyle. This condition further reduces their exercise capacity. In the literature, several studies have assessed the exercise capacity of these patients; however, these studies have predominantly utilized treadmill or cycle ergometers to evaluate lower extremity exercise capacity, and no study has been found that specifically investigates upper extremity exercise capacity. Considering that the upper extremities are used more frequently than the lower extremities during daily living activities, it is of particular importance to evaluate the upper extremity exercise capacity of patients. Moreover, upper extremity exercise testing provides an alternative means of assessment for patients with coronary artery disease who are unable to participate in lower extremity exercise tests due to neurological, vascular, or orthopedic problems. Compared to the lower extremities, the active muscle groups engaged during upper extremity exercise testing are smaller, which leads to lower metabolic demand and reduced peak oxygen consumption. This results in a lower cardiopulmonary workload during the exercise test. Therefore, it is necessary to investigate and compare upper and lower extremity exercise capacities, as well as the physiological responses elicited during exercise testing, in patients with coronary artery disease.

The primary aim of the study is to compare upper and lower extremity exercise capacities and arterial stiffness levels during exercise testing in patients with coronary artery disease.

The secondary aim of the study is to evaluate muscle oxygenation, energy expenditure, and the perception of dyspnea and fatigue during upper and lower extremity exercise testing in patients with coronary artery disease.

The primary outcomes are upper and lower maximal exercise capacities (Cardiopulmonary exercise tests) and arterial stiffness during cardiopulmonary exercise tests (Arteriograph) device).

Secondary outcomes are muscle oxygenation (Near-infrared spectroscopy) device, respiratory muscle fatigue (mouth pressure device), energy consumption (multi sensor activity device), the perception of dyspnea (Modified Borg Scale (MBS)) and fatigue (MBS).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-85 with coronary artery disease diagnosed by conventional or CT angiography
* Clinically stable
* Willing to participate

Exclusion Criteria:

* Heart failure diagnosis
* Moderate/severe valvular heart disease
* Orthopedic, neurological, or pulmonary conditions limiting exercise testing/capacity
* Contraindications per ACSM guidelines
* Prior coronary artery bypass graft surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients diagnosed with coronary artery disease will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Maximal Exercise Capacity | Through study completion, an average of 1 year
  Maximal Exercise capacity will be evaluated with Cardiopulmonary Exercise testing. The Cardiopulmonary Exercise Testing will be applied according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Arterial Stiffness [carotid-femoral pulse wave velocity (PWV)] | Through study completion, an average of 1 year
  Arterial stiffness will be non-invasively evaluated with using the SphygmoCor XCEL® device, which has established validity and reliability. The device will measure carotid-femoral pulse wave velocity (PWV) along with pulse values.
Arterial Stiffness [augmentation index (AIx)] | Through study completion, an average of 1 year
  Arterial stiffness will be non-invasively evaluated with using the SphygmoCor XCEL® device, which has established validity and reliability. The device will measure augmentation index (AIx) along with pulse values.

SECONDARY OUTCOMES:
Peripheral Muscle Oxygenation | Through study completion, an average of 1 year
  Peripheral muscle oxygen will be measured by near-infrared spectrometry. The device probes will be placed on the upper, lower extremities and trunk for both tests. The device allows to display of the percentage of oxygen, the concentration of oxyhemoglobin, and deoxyhemoglobin, the difference between oxyhemoglobin and deoxyhemoglobin, and the total hemoglobin. These parameters will be evaluated in our study.
Energy Consumption | Through study completion, an average of 1 year
  Energy consumption will be evaluated with the Multi sensor activity monitor. The patient wear the multi sensor physical activity monitor over the triceps muscle of the non-dominant arm during CPETs. Energy consumption (joule / day) will be measured with the multi-sensor physical activity monitor.
Peripheral Muscle Strength | Through study completion, an average of 1 year
  Isometric peripheral muscle strength will be measured with a portable hand dynamometer. Measurements will be repeated on the shoulder abductors and knee extensors three times on the right and left.
Respiratory Muscle Strength | Through study completion, an average of 1 year
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength were measured using a portable mouth pressure measuring device according to ATS and ERS criteria.
Respiratory Muscle Fatigue | Through study completion, an average of 1 year
  Respiratory muscle fatigue in patients will be assessed both before and immediately after upper and lower extremity cardiopulmonary exercise testing by measuring maximal inspiratory pressure (MIP) using a mouth pressure measurement device in accordance with ATS/ERS criteria. Prior to the tests, measurements will be repeated at least five times until the difference between the two highest MIP values is less than 5% or 5 cmH₂O. Immediately after the tests, at least three measurements will be performed until the difference between the two best MIP values is less than 5% or 5 cmH₂O.
Pulmonary Function (Forced vital capacity (FVC)) | Through study completion, an average of 1 year
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, forced vital capacity (FVC)was evaluated.
Pulmonary Function (Forced expiratory volume in first second (FEV1)) | Through study completion, an average of 1 year
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, forced expiratory volume in first second (FEV1) was evaluated.
Pulmonary Function (FEV1/FVC) | Through study completion, an average of 1 year
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, FEV1/FVC was evaluated.
Pulmonary Function (Flow rate 25-75% of forced expiratory volume (FEF25-75%)) | Through study completion, an average of 1 year
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, Flow rate 25-75% of forced expiratory volume (FEF25-75%)was evaluated.
Pulmonary Function (Peak flow rate (PEF)) | Through study completion, an average of 1 year
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, peak flow rate (PEF) was evaluated.
Physical Activity Level | Through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor. The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Physical activity level will be measured with the multi-sensor physical activity monitor.
Chronotropic Response Assessment | Through study completion, an average of 1 year
  Chronotropic response assessment will be evaluated through exercise testing using the chronotropic index, which is calculated based on the maximal heart rate achieved during the exercise test and the resting heart rate.
Dyspnea Perception | Through study completion, an average of 1 year
  Dyspnea perception will be evaluated with Modified Borg Scale. The Modified Borg scale is a subjective scale that scores 0-10 for breathlessness and fatigue at rest and/or during activity. The lowest 0 points "not at all" the highest 10 points "very severe" means shortness of breath.
Fatigue Perception | Through study completion, an average of 1 year
  Fatigue perception will be evaluated with Modified Borg Scale. The Modified Borg scale is a subjective scale that scores 0-10 for breathlessness and fatigue at rest and/or during activity. The lowest 0 points "not at all" the highest 10 points "very severe" means fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye SEVİM, Pt., Study Chair — Gazi University; Özden SEÇKİN, Dr., Principal Investigator — Gazi University; Mehmet Rıdvan YALÇIN, Prof.Dr., Principal Investigator — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya 06490, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442
- [Background] Secher NH, Volianitis S. Are the arms and legs in competition for cardiac output? Med Sci Sports Exerc. 2006 Oct;38(10):1797-803. doi: 10.1249/01.mss.0000230343.64000.ac. PMID 17019302
- [Background] Ranadive SM, Fahs CA, Yan H, Rossow LM, Agiovlasitis S, Fernhall B. Comparison of the acute impact of maximal arm and leg aerobic exercise on arterial stiffness. Eur J Appl Physiol. 2012 Jul;112(7):2631-5. doi: 10.1007/s00421-011-2238-z. Epub 2011 Nov 15. PMID 22083536
- [Background] Miles DS, Cox MH, Bomze JP. Cardiovascular responses to upper body exercise in normals and cardiac patients. Med Sci Sports Exerc. 1989 Oct;21(5 Suppl):S126-31. PMID 2691824
- [Background] Ghroubi S, Chaari M, Elleuch H, Massmoudi K, Abdenadher M, Trabelssi I, Akrout M, Feki H, Frikha I, Dammak J, Kammoun S, Zouari N, Elleuch MH. The isokinetic assessment of peripheral muscle function in patients with coronary artery disease: correlations with cardiorespiratory capacity. Ann Readapt Med Phys. 2007 Jun;50(5):295-301; 287-94. doi: 10.1016/j.annrmp.2007.03.012. Epub 2007 Mar 30. English, French. PMID 17449129
- [Background] Cakal B, Yildirim M, Emren SV. Kinesiophobia, physical performance, and health-related quality of life in patients with coronary artery disease. Postepy Kardiol Interwencyjnej. 2022 Sep;18(3):246-254. doi: 10.5114/aic.2022.122892. Epub 2022 Dec 17. PMID 36751297
- [Background] Alves AJ, Oliveira NL, Lopes S, Ruescas-Nicolau MA, Teixeira M, Oliveira J, Ribeiro F. Arterial Stiffness is Related to Impaired Exercise Capacity in Patients With Coronary Artery Disease and History of Myocardial Infarction. Heart Lung Circ. 2019 Nov;28(11):1614-1621. doi: 10.1016/j.hlc.2018.08.023. Epub 2018 Sep 19. PMID 30318391
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200